CLINICAL TRIAL: NCT01574560
Title: Community Outreach and Biomarker Feedback for Smoke-Free Homes
Brief Title: P60 Program Project Grant-Outreach for Smoke-Free Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2009NTLS058
Record Dates: First submitted 2012-04-05; First posted 2012-04-10 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Smoking Cessation; Tobacco Cessation
Keywords: smoke-free; tobacco exposure; biomarker feedback; nicotine; cotinine; secondhand smoke
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group - Health Education (Active Comparator): This group is provided with information regarding secondhand smoke and creating a healthy home environment.
  Interventions: Behavioral: Brochure
- Treatment Group - Counseling (Active Comparator): This group is provided with biomarker feedback on child exposure to secondhand smoke. Active participants receive 5 counseling sessions from a trained research counselor; 3 sessions in the home and 2 by phone. The counseling sessions focus on changing smoking behaviors and/or other behaviors that impact smoking.
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Brochure — Information regarding secondhand smoke and creating a healthy home environment.
  Arms: Control Group - Health Education
Behavioral: Counseling — Receives brochure and counseling sessions focusing on changing smoking behaviors and/or other health behaviors.
  Arms: Treatment Group - Counseling

SUMMARY:
Smoking is widely accepted to cause an increase in an individual's likelihood of developing cancer and heart disease. The effects of tobacco smoke are not limited to smokers. Secondhand smoke inhaled by a non-smoker has also been associated with the development of several illnesses. This study focuses on learning how to make your home smoke-free.

DETAILED DESCRIPTION:
This study will be conducted in two phases. Phase 1 will be qualitative focus groups/pilot study with the purpose to develop a motivationally enhanced biomarker feedback counseling protocol and all printed materials to be used in Phase 2. After investigators develop a good working treatment protocol, an active intervention in smoking homes who live with a child in their home will be carried out.

Those randomized to the Control Group will receive health education in the form of brochures detailing the health effects of secondhand smoke and how to make their home smoke free. Participants randomized to the Treatment Group will receive tobacco-specific biomarker feedback and personalized motivationally enhanced counseling.

ELIGIBILITY:
Inclusion Criteria (adult):

* Age 18 years or older
* Female
* Smoked ≥ 1 cigarettes per day for at least the past 6 months
* Smoked on 20 days or more in the last month
* Smoking status confirmed via cotinine verification strips
* Resides with a child ≤ 10 years of age in the role of the child's parent or caregiver
* Will agree to provide a urine sample at study enrollment
* Will also agree to the child providing a urine sample at study enrollment and at follow-up visits (for children who are not toilet trained, a diaper sample will be collected in lieu of the urine sample)
* Has a home address
* Has a functioning home phone or cell phone
* Provides written informed consent

Inclusion criteria (child):

* < or = 10 years of age
* Non-smoker -no cigarette use within prior 30 days to enrollment; however experimentation with smoking (a puff) will not exclude the child
* Lives in the primary home with the adult study participant at least 5 days a week

Exclusion criteria (adult):

* Current or past 7 day use of Nicotine Replacement Therapy (NRT) or pharmacotherapy for smoking cessation
* Planning to move outside of Minnesota within the next 3 months
* Have complete home smoking restrictions currently in place verified by the nicotine dosimeter
* Currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in Home Secondhand Smoke levels | From Baseline to Week 26 Follow-Up
  Measured by nicotine dosimeter - a passive "badge" hung in the home that measures free floating airborne nicotine particles.

SECONDARY OUTCOMES:
Comparison of Child Cotinine Levels in Urine | From Baseline to Week 26 Follow-Up
  Cotinine is an alkaloid found in tobacco and is also a metabolite of nicotine. Cotinine is used as a biomarker for exposure to tobacco smoke. Child (non-smoker) cotinine will be used as an objective measure of secondhand smoke exposure at baseline and again at end of study (week 26).
Comparison of Questionnaire Results | Baseline, Week 16 and Week 26
  Measured by mediators and moderators of effect, including psychosocial and tobacco-related variables.

CONTACTS AND LOCATIONS:
Overall Officials: Janet L. Thomas, Ph.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States